CLINICAL TRIAL: NCT03910322
Title: The Effect of Daily Intake of Two Different Doses of Bif195 on Small-intestinal Damage Induced by Acetylsalicylic Acid- a Randomized, Double-blind, Placebo-controlled, Three-armed, Parallel Group Trial in Healthy Volunteers.
Brief Title: The Effect of a Probiotic Strain on Aspirin-induced GI Damage
Acronym: PIP-L
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made by Sponsor
Sponsor: Chr Hansen (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-GI-035
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2019-08

CONDITIONS: Reduction of Small Intestinal Ulceration Risk

STUDY DESIGN:
Intervention Model Description: This trial is a single-site, randomized, double-blind, placebo-controlled, three-armed, parallel-group trial in healthy volunteers aged 40 - 60 years. The trial will investigate the effect of daily intake of the probiotic strain Bif195 in two different doses or placebo when co-administered to daily intake of 300mg of Acetylsalicylic Acid (ASA).
  The trial includes a run-in period of two weeks duration followed by a six weeks intervention period where Bif195/placebo and ASA is co-administered.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo arm. Similar trial product, but without Bif195 bacteria
  Interventions: Dietary Supplement: Placebo
- Low-dose Bif195 (Experimental): Active trial product with minimum 15 billion CFU daily dose
  Interventions: Dietary Supplement: Bif195
- High-dose Bif195 (Experimental): Active trial product with minimum 50 billion CFU daily dose
  Interventions: Dietary Supplement: Bif195

INTERVENTIONS:
Dietary Supplement: Bif195 — Two different doses of the bacterial strain Bif195 is compared to placebo
  Arms: High-dose Bif195; Low-dose Bif195
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate if a daily dose of minimum 50 billion CFU of Bif195 reduces the risk of small-intestinal tissue damage in an acetylsalicylic acid challenge model as assessed by video capsule endoscopy in a healthy US population aged 40 - 60 years.

DETAILED DESCRIPTION:
This trial is a single-site, randomized, double-blind, placebo-controlled, three-armed, parallel-group trial in healthy volunteers aged 40 - 60 years. The trial will investigate the effect of daily intake of the probiotic strain Bif195 in two different doses or placebo when co-administered to daily intake of 300mg of Acetylsalicylic Acid (ASA).

The trial includes a run-in period of two weeks duration followed by a six weeks intervention period where Bif195/placebo and ASA is co-administered.

Subjects will participate in the trial for a total duration of 8 weeks including the run-in phase. Besides the screening visit, the trial will consist of 5 visits.

After having given their written informed consent, subjects will complete the screening procedures to evaluate their eligibility for participation in the trial and complete a run-in period of two weeks duration to washout possible pre-trial probiotics and/or use of medication. After baseline assessments at Visit 2, subjects will start daily intake of 300mg ASA and also be randomly assigned to 6-weeks daily intake of low or high-dose active (Bif195) or placebo product in a ratio of 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy and without any gastrointestinal discomfort/pain symptoms
* Age 40-60 years of both genders (aim of minimum 1/3 of each gender in each arm)
* Willing and able to abstain from any other probiotic products and/or medication known to alter gastrointestinal function throughout the participation of the trial

Exclusion Criteria:

* Abdominal surgery which, as judged by the investigator, might affect the GI function (except appendectomy and cholecystectomy)
* History of peptic ulcer disease
* Any known bleeding disorder
* Allergy to ASA
* Resting diastolic blood pressure ≥ 95 mmHg
* Resting systolic blood pressure ≥ 150 mmHg
* A current diagnosis of psychiatric disease
* Systemic use of antibiotics, steroids (except contraceptives) or antimicrobial medication in the last 2 months
* Daily usage of non-steroidal anti-inflammatory drugs in the last 2 months or incidental use in the last 2 weeks prior to screening (ASA, Ibuprofen, Diclofenac, Naproxen, Celecoxib, Mefenamic acid, Etoricoxib, Indometacin)
* Usage of medications, except contraceptives, in the last 2 weeks prior to screening
* Diagnosed inflammatory gastrointestinal disease and/or irritable bowel syndrome
* Any other disease that, by the Investigators discretion, could interfere with the intestinal barrier function of the subject
* Participation in other clinical trials in the past 2 months prior to screening
* Regular use of probiotics in the last month
* Smoking and/or frequent use of other nicotine products
* Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial
* Use of laxatives, anti-diarrheals, anti-cholinergics and proton pump inhibitors within last 2 months prior to screening
* Use of immunosuppressant drugs within last 4 weeks prior to screening
* For Women: Pregnancy or lactation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
primary endpoint - Lewis score high dose Bif195 vs Placebo | 6 weeks
  The effect of high-dose Bif195 versus placebo on small intestinal mucosal damage during a 6-week ASA challenge measured as the area-under-the-curve of the Lewis scores obtained from all video capsule endoscopies between Visit 2 (randomization) and Visit 6 (end of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Eamonn Quigley, Professor, Principal Investigator — Houston Methodist Gastroenterology Associates
Locations (1):
- Atlantia Food Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No